CLINICAL TRIAL: NCT00203333
Title: Cardiac Rhythm Abnormalities in Patients With Refractory Epilepsy at High Risk for Sudden Death
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: J05901
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Refractory Epilepsy; Arrhythmia; Sudden Death
Keywords: Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy; Arrhythmias, Cardiac; Death, Sudden; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Medtronic REVEAL

SUMMARY:
People with epilepsy are at a higher risk for sudden unexpected death than the general population. Sudden unexpected death in epilepsy (SUDEP) is a major cause of death in this population, accounting for 10-50% of deaths for those with epilepsy. The risk for SUDEP is particularly high for those with refractory epilepsy. Several lines of evidence support a cardiac mechanism for SUDEP.

This study plans to determine:

1. the frequency and types of cardiac arrhythmias that occur in this population and
2. whether these are increased above the general population in the same age group.

Additionally, these data will be correlated to specific clinical data, including seizure history, anticonvulsant medications, and any accompanying clinical symptoms.

DETAILED DESCRIPTION:
By employing long-term electrocardiographic monitoring, this study plans to determine:

1. the frequency and types of cardiac arrhythmias that occur in patients with uncontrolled seizures and
2. whether these are increased above the general population in the same age group.

The specific aims:

1. Identify the types, frequency, and duration of cardiac arrhythmias that occur in patients with refractory epilepsy and compare these data to available normative data.
2. Correlate abnormal heart rates and rhythms to specific clinical data:

   1. seizure type,
   2. seizure frequency,
   3. probable location of seizure onset in the brain, when such data are available,
   4. duration of seizures, and
   5. type(s) and number of anticonvulsant medications being used.
3. Correlate cardiac arrhythmias to clinical symptoms

ELIGIBILITY:
Inclusion Criteria:

* Refractory epilepsy

Exclusion Criteria:

* Other pre-existing heart conditions

Ages: 16 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals with refractory focal or generalized epilepsy.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2002-04; Primary Completion 2007-06 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maromi Nei, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Nei M, Sperling MR, Mintzer S, Ho RT. Long-term cardiac rhythm and repolarization abnormalities in refractory focal and generalized epilepsy. Epilepsia. 2012 Aug;53(8):e137-40. doi: 10.1111/j.1528-1167.2012.03561.x. Epub 2012 Jun 18. PMID 22709423